CLINICAL TRIAL: NCT00867178
Title: A Feasibility Study of Vorinostat (SAHA) Combined With Isotretinoin and Chemotherapy in Infants With Embryonal Tumors of the Central Nervous System
Brief Title: Vorinostat Combined With Isotretinoin and Chemotherapy in Treating Younger Patients With Embryonal Tumors of the Central Nervous System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03167; NCI-2012-03167 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-026; PBTC-026 (Other: Pediatric Brain Tumor Consortium); PBTC-026 (Other: CTEP); U01CA081457 (NIH); UM1CA081457 (NIH)
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-09

CONDITIONS: Medulloblastoma; Pineoblastoma; Supratentorial Embryonal Tumor, Not Otherwise Specified
MeSH Terms: conditions — Medulloblastoma; Pinealoma | interventions — Radiotherapy, Conformal; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; etoposide phosphate; Isotretinoin; Peripheral Blood Stem Cell Transplantation; Thiotepa; Vincristine; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (vorinostat, isotretinoin, chemotherapy) (Experimental): See Detailed Description
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Etoposide Phosphate; Drug: Isotretinoin; Other: Laboratory Biomarker Analysis; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Thiotepa; Drug: Vincristine Sulfate; Drug: Vorinostat

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo conformal radiation therapy
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
Drug: Isotretinoin — Given PO
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Absorica; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Myorisan; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret; ZENATANE
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSC
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This pilot clinical trial studies the side effects and the best way to give vorinostat with isotretinoin and combination chemotherapy and to see how well they work in treating younger patients with embryonal tumors of the central nervous system. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as isotretinoin, vincristine sulfate, cisplatin, cyclophosphamide, and etoposide phosphate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving vorinostat with isotretinoin and combination chemotherapy may be an effective treatment for embryonal tumors of the central nervous system. A peripheral blood stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. This may allow more chemotherapy to be given so that more tumor cells are killed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the feasibility of administering vorinostat (SAHA) and isotretinoin for three days prior and concomitant with cisplatin based chemotherapy over three courses of induction chemotherapy.

II. To describe the toxicity of administering vorinostat (SAHA) and isotretinoin for three days prior and concomitant with cisplatin based chemotherapy over three courses of induction chemotherapy.

III. To investigate prognostic values of histopathological classification and biological markers in the context of a feasibility study.

SECONDARY OBJECTIVES:

I. To estimate the preliminary response rate of this approach in patients with measurable residual disease (primary site and/or metastatic sites).

II. To estimate disease specific progression-free and overall survival, in the context of a feasibility study.

III. To explore the predictive values of biological markers in cerebrospinal fluid (CSF), plasma, urine tumor material in the context of a feasibility study.

OUTLINE:

INDUCTION THERAPY: Patients receive vorinostat orally (PO) once daily (QD) and isotretinoin PO twice daily (BID) on days 1-4; vincristine sulfate intravenously (IV) on days 4, 11, and 18; cisplatin IV over 6 hours on day 4; cyclophosphamide IV over 1 hour on days 5-6; and etoposide phosphate IV over 1 hour on days 4-6. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo peripheral blood stem cell (PBSC) harvesting after each course.

CONSOLIDATION THERAPY: Within 6 weeks (10 weeks if patient is re-staged) after completion of induction therapy, patients receive carboplatin IV over 2 hours and thiotepa IV over 2 hours on days 1-2. Patients also receive autologous PBSC rescue infusion over 6 hours on day 4. Treatment repeats every 28 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Beginning 3 weeks later, patients with M0 non-desmoplastic medulloblastoma also undergo conformal radiotherapy* to the tumor bed.

NOTE: *Patients with supratentorial primary tumors or metastatic disease undergo radiotherapy at the discretion of treating physician.

MAINTENANCE THERAPY: Beginning 4 weeks after completion of radiotherapy or immediately after completion of consolidation therapy, patients receive vorinostat PO QD on days 1, 3, 5, 6, 8, 10, 12, and 13 and isotretinoin PO BID on days 1-14. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed, newly-diagnosed medulloblastoma (except for patients with the histology of localized (M0) desmoplastic medulloblastoma or atypical teratoid/rhabdoid tumor [ATRT]) or supratentorial primitive neuroectodermal tumor (PNET) including pineoblastomas
* Patients must have not received any prior therapy other than surgery and/or steroids
* Patient must have adequate pre-trial formalin-fixed, paraffin-embedded (FFPE) tumor material available for use in the biology studies and central pathology review; if snap frozen tissue is not available, the study chair must be contacted to discuss eligibility
* Patient must be a suitable candidate, by institutional standards for stem cell apheresis
* Lansky performance score (LPS for =< 16 years of age) >= 30 assessed within two weeks prior to registration
* Absolute neutrophil count (ANC) >= 1000/ul (unsupported) (within 14 days of registration and within 7 days of the start of treatment)
* Platelets >= 100,000/ul (unsupported) (within 14 days of registration and within 7 days of the start of treatment)
* Hemoglobin >= 8 g/dL (may be supported) (within 14 days of registration and within 7 days of the start of treatment)
* Bilirubin < 1.5 times upper limit of normal for age (within 14 days of registration and within 7 days of the start of treatment)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 1.5 times institutional upper limit of normal for age (within 14 days of registration and within 7 days of the start of treatment)
* Serum creatinine =< 1.5 times upper limit of institutional normal for age or glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or estimated GFR (Schwartz bedside) that is > 99 ml/min/1.73 m^2 (within 14 days of registration and within 7 days of the start of treatment)
* Parents/legal guardians must have the ability to understand and the willingness to sign a written informed consent document according to institutional guidelines

Exclusion Criteria:

* Patients with diagnosis of atypical teratoid/rhabdoid tumor (ATRT by histology, immunohistochemistry and/or molecular analysis) and desmoplastic M0 medulloblastoma will be excluded from the study
* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that would compromise the patient's ability to tolerate protocol therapy or would interfere with the study procedures or results
* Patients receiving any other anticancer or investigational drug therapy are excluded
* Patients having taken valproic acid within 2 weeks prior to initiation of treatment are excluded
* Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy
* Patients with a parabens allergy

Ages: 2 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2009-02-25 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity of proposed vorinostat | Up to 21 days
  Will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Feasibility in terms of completing 3 courses of induction therapy | Within 98 days
  Simon's two-stage optimal design will be used to assess feasibility.
Prognostic value of histopathological classification of pediatric medulloblastoma | Up to 5 years
  Will be assessed by single-nucleotide polymorphism (SNP) analysis and gene expression analysis. Loss of heterozygosity (LOH) analysis and copy number analysis (CNA) will be performed using dChip SNP software (or R bioconductor package) for the paired samples. Association of copy number (and LOH) with gene expression data will be explored. Correlation analysis (Pearson or Spearman Correlation, as appropriate) will be used to estimate the strength of association between each SNP and expression signal. The multiplicity issue will be addressed through estimating the False Discovery Rate.

SECONDARY OUTCOMES:
Response rate of this approach in patients with measurable residual disease (primary site and/or metastatic sites) | Up to 5 years
  Separate exact confidence interval estimates of objective responses following induction therapy will be constructed for patients with medulloblastomas (MBs) and PNETs. Cumulative incidence of objective responses as a function of course of therapy will also be provided.
Progression-free survival (PFS) | Up to 5 years
  Kaplan-Meier estimates of distributions of PFS will be provided. If sample sizes allow, these Kaplan-Meier estimates will be produced separately for patients with MBs and PNETs.
Overall survival (OS) | Up to 5 years
  Kaplan-Meier estimates of distributions of OS will be provided. If sample sizes allow, these Kaplan-Meier estimates will be produced separately for patients with MBs and PNETs.
Predictive values of biological markers in CSF, plasma and urine in the context of a feasibility study | Up to 5 years
  Frequency of the markers of interest present in this cohort will be provided and their associations with disease outcome will be explored. Similarly if sample size constraints make such analyses feasible, the associations between the markers of interest and clinical and demographic variables will be explored in a descriptive fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Leary, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (15):
- United States (15):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - National Cancer Institute Pediatric Oncology Branch, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Pediatric Brain Tumor Consortium, Memphis, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington